CLINICAL TRIAL: NCT05858476
Title: An Investigation Into a 21-Day Detoxification Diet With a Seven-Day Continuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chef V, LLC (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20267
Record Dates: First submitted 2023-04-22; First posted 2023-05-15 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2023-05

CONDITIONS: Detoxification
MeSH Terms: interventions — detox adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chef V's 21-Day Starter Challenge Detox & Green Drink Supplement (Experimental): The detox program provides the three primary macronutrients alongside antioxidants to promote detoxification. The 21-Day Detox schedule is below:
  Days 1-7: Healthy Routine- The Healthy Routine involves drinking a 16oz Green Drink and Protein Shake for breakfast and then choosing their lunch, snack, and dinner from the Meal Planner that will be provided.
  Days 8-10: 3-Day Cleanse- Each day during the three-day cleanse, participants will consume 4 16oz Green Drinks, 2 Protein Shakes, and a Soup designed explicitly to detox the body.
  Days 11-21: Healthy Routine- The last period of the 21 days will mimic the Healthy Routine from Days 1-7.
  Days 21-28 Participants will follow up this program by using the Green Drink supplement provided for an additional 7 days.
  Interventions: Other: 21-Day Detox and Green Drink supplement

INTERVENTIONS:
Other: 21-Day Detox and Green Drink supplement — Detox plan description:
  7AM Water 16oz. 8AM Green Drink 16oz. 9AM Ultra Shake 16oz. 9-12PM Water 24 - 48oz. 12PM Green Drink 16oz. 12:30 - 2PM Water 24 - 48oz. 2PM Green Drink 16oz. 3PM Ultra Shake 16oz. 3:30- 6PM Water 24 - 48oz. 6PM Green Drink 16oz. 7PM Detox Soup 16oz. 7:30 - 10PM Water 24 - 48oz. This 21-day period will be followed by 7 days of consuming the Green Drink Supplement.

SUMMARY:
Detoxification diets aim to remove chemicals from the body that may cause short or long-term harm. However, little is known about detoxification diets from well-designed clinical trials. This trial examines the efficacy of Chef V's 21-Day Starter Challenge Detox diet. Participants will use Chef V's 21-Day Starter Challenge Detox as directed for the first 21 days of the trial and continue to use the Chef V Green Drink Supplement for an additional seven days. The primary outcomes of interest are the participant's perceptions of their health improvements and biomarkers that will be measured via blood draws.

ELIGIBILITY:
Inclusion Criteria:

* Must be in good general health with no chronic health conditions
* BMI under 35.
* Must own a scale at home.
* Must experience at least one of the following issues: the feeling of being tired at least several times a week, brain fog, sleep issues, trouble with focus and concentration, or having a busy, stressful life.
* A subgroup of 10 study participants must be diagnosed with T2D for ≥ 90 days, with an hbA1c of 7.5 to 10.5, inclusive
* Eat fast food at least twice a week.
* Does not exercise regularly.
* Does not consume fruits and vegetables daily.
* Must experience at least one of the following gastrointestinal problems: often bloating, excessive gas, heartburn, and irregular bowel movements.
* Must experience at least one of the following aches regularly: body aches, joint pain, back pain, or neck pain.
* Must be willing to go to Quest labs for two blood draws, one at baseline and the other at the study's conclusion.
* Willing to avoid bottled water for the duration of the study.

Exclusion Criteria:

* Suffers from pre-existing conditions that prevent them from adhering to the protocol.
* Anyone with known severe allergic reactions.
* Currently pregnant, breastfeeding, or wanting to become pregnant for the duration of the study.
* Anyone unwilling to use the test product daily as directed.

Ages: 31 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2022-12-02 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Changes in participant perceptions of well-being [Time Frame: Baseline to 28 days) | 28 days
  Survey-based assessment (0-5 scale) of changes in IBS symptoms). Participants will answer surveys at the study baseline, and on Days 5, 11, 21 and 28 of the trial.

SECONDARY OUTCOMES:
Change in hs-CRP [Time Frame: Baseline to 28 days] | 28 days
  Blood draws will be taken at Baseline and Day 28 for comparison.
Change in blood lipid profile [Time Frame: Baseline to 28 days] | 28 days
  Blood draws will be taken at Baseline and Day 28 for comparison.
Change in HbA1C [Time Frame: Baseline to 28 days] | 28 days
  Blood draws will be taken at Baseline and Day 28 for comparison.
Change in bodyweight [Time Frame: Baseline to 28 days] | 28 days
  Weight will be measured using an electric scales at the study baseline and on Days 3, 5, 14, and 18.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States